CLINICAL TRIAL: NCT06176833
Title: Critical Time Window for Rehabilitation After Incomplete Spinal Cord Injury: Early vs Late Locomotor Training
Brief Title: Promoting Recovery Outcomes Through Precise Early Locomotor Interventions in Persons With Spinal Cord Injury
Acronym: PROPEL-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milap Sandhu (Other)
Collaborators: Baylor Scott and White Health (Other); University of Florida (Other)
Responsible Party: Sponsor-Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00219541
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of 4 intervention groups, based around if and when additional walking training is given following injury
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will have no knowledge of groups, cannot blind participants as they know when they will be receiving the additional training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Intervention (Active Comparator): Additional training will begin no more than 60 days following spinal cord injury
  Interventions: Procedure: Body Weight Supported Treadmill Training
- Sub-acute Intervention (Active Comparator): Additional training will occur 3 months following spinal cord injury
  Interventions: Procedure: Body Weight Supported Treadmill Training
- Chronic Intervention (Active Comparator): Additional training will occur 6-12 months following SCI
  Interventions: Procedure: Body Weight Supported Treadmill Training
- Standard of Care (No Intervention): This group only receives standard of care treatment but is assessed at the same time points as the other groups

INTERVENTIONS:
Procedure: Body Weight Supported Treadmill Training — For these training sessions, participants will undergo walking training sessions that consist of wearing a harness for either body weight support or as a safety precaution while walking on a treadmill.
  Other Names: BWSTT
  Arms: Chronic Intervention; Early Intervention; Sub-acute Intervention

SUMMARY:
The purpose of this study is to evaluate if a specific type of additional walking therapy, called body weight supported treadmill training (BWSTT) affects walking ability following a traumatic spinal cord injury. Specifically, the study will look at whether starting BWSTT, which uses a body harness to support body weight while walking on a treadmill at different times within the first 6 months after the injury, makes a difference in how effective this therapy may be, While we know that the brain re-learns patterns following an injury, there has not been a lot of prior research evaluating how starting this type of walking therapy at specific times within the first 6 months after injury may impact any effectiveness of the additional therapy.

The study will randomize participants into four groups: those who start this therapy within 60 days, within 3 months, within 6 months or who do not receive this additional research therapy. Randomization means that which group you will be in as part of this study is determined by chance, like the flip of a coin. The additional walking therapy for this research study, if you are randomized for one of the three groups who receives the additional therapy, will be given on top of (meaning in addition to) any standard of care therapies that you may be receiving at that time point after your injury.

ELIGIBILITY:
Inclusion Criteria:

* History of Acute and Traumatic SCI with AIS classification of B, C, or D between the neurological levels of C5 and T12
* Between the ages of 16-74
* Weight bearing as tolerated in bilateral lower extremities
* Able to tolerate a harness
* Ability to provide informed consent. For minors, consent of parents or primary caregivers/guardians and assent of the minor
* Able to provide informed consent within 60 days of injury onset
* Able to participate in all study related activities, including 1-year follow up

Exclusion Criteria:

* Orthopedic injuries, fractures, surgeries, or other conditions affecting locomotor function or weight bearing
* A weight over 250lbs and if so a BMI greater than 30, or deemed clinically inappropriate due to body habitus
* Moderate to sever traumatic brain injury of other neurological conditions at a severity which impairs cognition
* Presence of uncontrolled orthostatic hypotension that limits active participation in intense physical rehabilitation program.
* Other medical complications such as severe heart failure or large/deep pelvic or lower abdominal wounds that may limit the ability to safely don and doff a harness for ambulation
* Pregnancy, as confirmed by blood draw

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
10 Meter walk test | 1-5 days Following Intervention
  Used to assess walking speed, time taken to walk 10 meters at fastest pace

SECONDARY OUTCOMES:
6 Minute Walk test | 1-5 days Following Intervention
  Used to assess distance traveled during a 6 minute walking test at a self selected pace
Walking Index for spinal cord injury | 1-5 days following intervention
  Assessment to determine the physical assistance and assistive devices needed to walk 10 meters
Daily step counts | 2 weeks following 3-, 6-, 9-, and 12- month assessments
  Step counts from a waist worn activity tracker
Gait Deviation idex | Baseline, 3-, 6-, 9-, and 12- month assessments
  A measure of gait quality by quantifying joint angles during a gait cycle. This data is recorded via a marker-less motion capture system

CONTACTS AND LOCATIONS:
Overall Officials: Milap Sandhu, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - The Shirley Ryan AbilityLab, Chicago, Illinois
  - Baylor Scott and White Institute for Rehabilitation, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
We are not currently planning to make individual participant data available to other researchers

REFERENCES:
- [Derived] Henry M, Coxe RC, Barry A, O'Donnell A, Kessler A, Shan G, Swank C, Rymer WZ, Sandhu MS. A research protocol to study the critical time window for rehabilitation after incomplete spinal cord injury: early vs. late locomotor training. BMC Neurol. 2024 Dec 19;24(1):482. doi: 10.1186/s12883-024-03980-x. PMID 39702102